CLINICAL TRIAL: NCT00644514
Title: The Genetics of Environmental Asthma: LPS Inhalation and Bronchoscopy in Normal Subjects and Subjects With Mild Atopic Asthma
Brief Title: Genetics of Asthma - Bronchoscopy Studies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: grant funding no longer available
Sponsor: John Sundy (Other)
Responsible Party: Sponsor-Investigator, John Sundy, Associate Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00001166; Pro00001166; 12496-CP-001A (Other: NIEHS)
Record Dates: First submitted 2008-03-24; First posted 2008-03-26 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: Atopic Asthma; Healthy
Keywords: LPS endotoxin; Asthma
MeSH Terms: conditions — Asthma | interventions — Lipopolysaccharides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LPS endotoxin inh f/u bronchoscopy (Experimental): Participants receive inhalation of LPS endotoxin, followed by bronchoscopy in this study.
  Interventions: Biological: Endotoxin - lipopolysaccharide (LPS)

INTERVENTIONS:
Biological: Endotoxin - lipopolysaccharide (LPS) — Nebulized 5000EU, 10,000EU, 20,000EU endotoxin doses delivered to completion. Nebulized dose inhaled 30 minutes apart if no adverse events occur after the previous dose. Fiberoptic Bronchoscopy with Bronchoalveolar Lavage (BAL) and brush samples performed 24 hours after LPS nebulization.
  Other Names: Lipopolysaccharide (LPS); NIH Clinical Center Reference Endotoxin

SUMMARY:
The purpose of this study is to identify the mediators and genes in airway epithelial and BAL cells that are differentially regulated following inhalation of endotoxin lipopolysaccharide (LPS) among study participants with allergic asthma and normal phenotypes. This approach is designed to identify novel genes associated with both asthma pathogenesis and asthma susceptibility. LPS, or endotoxin, a cell wall component of gram-negative bacteria, is ubiquitous in the environment, and is thought to influence both susceptibility and severity of asthma.

240 subjects (healthy adult men and women (age >18-40) with and without atopy and asthma) will complete the screening evaluations in order to establish 3 study groups of 60 subjects each. Each qualified subject will undergo an inhaled LPS endotoxin challenge followed by bronchoscopy after 24 hours, which will consist of a bronchoalveolar lavage (BAL) and endobronchial brush biopsies. BAL involves squirting a small amount of sterile salt water into one of the airways then gently taking it back out through the bronchoscope. The brush sample involves gently moving a small brush back and forth in an airway to collect cell samples. Samples of whole blood will also be obtained at various time points. RNA will be isolated from these cell populations in order to assess differential gene expression expression using microarrays.

DETAILED DESCRIPTION:
Background:

Endotoxin or lipopolysaccharide (LPS), a cell wall component of gram-negative bacteria, is ubiquitous in the environment, and is often present in high concentrations in organic dusts, as well as in air pollution, and household dusts. There is convincing evidence that endotoxin exacerbates airflow obstruction and airway inflammation in allergic asthmatics. Additional findings indicate that allergic airways can enhance the response to inhaled endotoxin, and that endotoxin can enhance the airway response to allergens. However, when considering the interaction between endotoxin and allergens, the timing of the exposure appears to be critical. Emerging evidence suggests that early exposure to endotoxin, a potent inducer of Th1 type cytokines (IFN-g and IL-12), may minimize the risk of allergen sensitization which could has profound effects on reducing the risk of developing asthma in children. Independent of its effect in allergic asthma, several studies demonstrate that inhalation of air contaminated with endotoxin is associated with the classical features of asthma (reversible airflow obstruction and airway inflammation, and persistent airway hyperreactivity and airway remodeling). Epidemiological studies have shown that the concentration of inhaled endotoxin in the bioaerosol is strongly and consistently associated with reversible airflow obstruction among cotton workers, agricultural workers, and fiberglass workers. Importantly, the concentration of endotoxin in the bioaerosol is the most important occupational exposure associated with the development and progression of airway disease in agricultural workers. Experimentally, inhalation of endotoxin can cause reversible airflow obstruction and airway inflammation in previously unexposed healthy study subjects. The ability of the host to respond to endotoxin is highly variable, and is influenced in part by genetic factors.:

The rationale for this investigation is based on the following points:

* asthma is caused in large part by both genetic susceptibility and environmental exposure,
* a variety of immune and non-immune mechanisms can function independently or interactively to cause airway hyper-reactivity, airflow obstruction, airway inflammation, and airway remodeling,
* environmental challenges can be used to "narrow the asthma phenotype" and allow one to investigate unique gene-environment interactions that are involved in the development of biologically specific forms of asthma,
* genes that are over or under stimulated in the airway epithelia of asthmatics following inhalation challenge are important in the pathogenesis of asthma

ELIGIBILITY:
Inclusion Criteria:

* Allergic asthmatic, allergic non-asthmatic, or nonallergic nonasthmatic
* Willing/able to give informed consent & adhere to visit/protocol schedules.
* Screening visit laboratory, C-Xray, EKG, results within normal limits
* Women of childbearing potential must have a negative serum pregnancy test
* Screening Pulmonary function testing above study criteria parameters

Exclusion Criteria:

* Systemic corticosteroid administration for asthma within the previous 90days
* Antibiotic administration within the previous 30 days.
* Viral respiratory infection within the previous 14 days.
* History of severe asthma requiring intubation.
* Occupational exposure to hay or grain dust.
* Significant exposure history to cigarette smoke
* Past or present history of allergen immunotherapy to within the last 10 yrs
* Underlying illnesses that may result in altered lung function
* Students or employees under direct supervision by protocol investigators are ineligible
* Subjects allergic to medications used (or potentially used) in the study will be excluded.
* Subjects using aspirin will be excluded
* Subjects who abuse alcohol or illicit substances will be excluded
* Medication use other than for asthma, allergies or contraception
* Other medical or psychological conditions which, in the opinion of the investigator, might create undue risk to the subject or interfere with the subject's ability to comply with the protocol requirements
* Nursing mothers
* Other investigational medication within the last 30 days

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2007-09; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Identify Genes in airway epithelial and Bronchoalveolar Lavage (BAL)that are differentially regulated following inhalation of LPS endotoxin. | bronchoscopy performed 24 hours after inhalation of endotoxin

SECONDARY OUTCOMES:
Identify mediators in airway epithelial and BAL cells that are differentially regulated following LPS inhalation. | Bronchoscopy performed 24 hours post inhalation of endotoxin

CONTACTS AND LOCATIONS:
Overall Officials: John S Sundy, M.D., PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States